CLINICAL TRIAL: NCT04153552
Title: Evaluation of the Impact of the HLNatural, Inc. Upset Stomach Relief Product on the Reduction of Symptoms in Adults Who Suffer From Mild to Moderate Indigestion and Heartburn
Brief Title: Upset Stomach Relief for Mild and Moderate Indigestion and Heartburn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawthorne Effect Inc. (Other)
Collaborators: HLNatural, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00037630
Record Dates: First submitted 2019-09-13; First posted 2019-11-06 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Indigestion; Heartburn
Keywords: Natural; Supplement
MeSH Terms: conditions — Dyspepsia; Heartburn

STUDY DESIGN:
Intervention Model Description: The present study will be a single site, prospective, one arm observational study of minimal risk consisting of at least 200 participants who suffer from symptoms of occasional indigestion and heartburn. Participants will begin taking the capsules at the onset of indigestion and heartburn symptoms. Onset is defined as the point in time the participant takes the test product for relief of symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants who Suffer from Heartburn or indigestion (Other): Subjects who meet the inclusion/exclusion criteria for the trial will be invited to participate in the trial. Subjects will be asked to sign a consent and complete screening survey. At the onset on an episode of the subject will start a symptom diary and completed and rate the symptoms using a 4-point Likert scale for each symptom. The participant will take 2 capsules per indigestion and heartburn episode. With a max of 6 capsules per day. • After taking the test product, the participant will complete a 4-point Likert scale assessment for each symptom at 15 minutes, 30 minutes, and 1 hour after taking the test product.
  Interventions: Dietary Supplement: HLNatural, Inc. Upset Stomach Relief

INTERVENTIONS:
Dietary Supplement: HLNatural, Inc. Upset Stomach Relief — Supplement to take with mild to moderate indigestion. The degree of your indigestion pre and post will be recorded

SUMMARY:
The primary hypothesis of the present study is that supplementation with the Upset Stomach Relief test product will reduce the severity of the symptoms of occasional indigestion and heartburn.

DETAILED DESCRIPTION:
The purpose of the present study is to evaluate 1) the impact of the test product on symptoms of occasional indigestion and heartburn in 200 adult participants who suffer from occasional indigestion and heartburn and 2) the subjective experience of these participants related to general health, indigestion and heartburn symptoms, and personal experience with the test product.

While dietary and lifestyle changes can ease the symptoms of indigestion and heartburn, HLNatural, Inc. created the test product to reduce occasional indigestion and heartburn. The test product is a plant-based remedy formulated with ingredients that have demonstrated efficacy reducing symptoms associated with occasional indigestion and heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Adult candidates who are in overall good health but who suffer from the symptoms of indigestion.
* Participants will be deemed to be in good health if they do not report any of the existing medical conditions asked about in the screening questionnaire.

Exclusion Criteria:

* Age <18 years old.
* Unwilling to take test product for their symptoms.
* Are not able to swallow pills.
* Allergy to any of the following: Licorice, Artichoke Leaf, Marshmallow Root, Ginger, Chamomile, Cellulose Capsule, Rice Hull Concentrate, Carrageenan.
* Has any of the following medical conditions:

  * Has had an ulcer
  * Has been diagnosed with a digestive disorder
  * Diagnosed with gastroesophageal reflux disorder
  * Participants with diagnosed with irritable bowel syndrome
  * Participants with active HP infection or with gastric or duodenal ulcer
* Participants who have been prescribed any medication by their physician for any GI disorder or medication that can affect the GI system.
* Participants with previous diagnosis of cancer or with previous surgery of the upper gastrointestinal tract or of the biliopancreatic system (except for cholecystectomy)
* Pregnant women or breastfeeding.
* Alcohol consumption more than 7 drinks per week or more than 3 drinks per occasion
* Participant who scores a 0, 3, or 4 on the Dyspepsia Symptom Severity Index
* Participants who are currently using anticoagulation medications daily. (Aspirin, Coumadin, Heparin etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 161 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Outcomes of the severity and reduction of indigestion while consuming HLNatural Supplement. | The improvements in symptoms will be evaluated from baseline.
  Participants will be asked to rate each symptom (bloating, early fullness during a meal, pain or discomfort in the upper abdomen, burning in the upper abdomen, pain/burning in the center of your chest, nausea, vomiting, and burping) on a 4-point scale at 4 time points. • At the onset of the indigestion and heartburn episode, the participant will start a Symptom Diary and complete a 4-point Likert scale for each of the symptoms they are experiencing.

SECONDARY OUTCOMES:
Outcomes of time to relief or to alternative treatment while taking HLNatural Supplement | The subject will write down symptoms in a diary and start of symptoms and again at 60 mins. The subject ill complete 4-point Likert Scale at start of event, 15 minutes, 30 minutes and 60 minutes after start of event.
  The participant is allowed to take alternative medications or supplements AFTER 1 hour from taking the test product. • If the participant takes any other medication outside of the test product, the participant will record this on the symptom diary.
Outcomes of all adverse events while consuming HLNatural Supplement | All adverse events will be captured throughout the trial which will be up to 60 days or 3 episodes of indigestion.
  Participants will be asked to report any adverse events that the subject experiences throughout the study.
Outcome of subjects natural behavior during the clinical trial | The time point will be evaluated from baseline to thoughout the trial up 60 days or 3 episodes of indigestion.
  At the start of the study participants will be asked to complete screening, baseline and demographic survey. At the completed of the study an exit study will be completed. This information along with what appears in the literature will help the investigators to better understand expected normal behavior of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Soyona Rafatjah, MD, Principal Investigator — Hawthorne Effect Inc.
Locations (1):
- HLNatural, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once the trial is completed and the data has been analyzed then a decision will be made on how to use the data.

REFERENCES:
- [Background] 1. 15 Pain Scales (And How to Find The Best Pain Scale For You). (2018, January 05). Retrieved from https://paindoctor.com/pain-scales/
- [Background] 2. Artichoke: Uses, Side Effects, Interactions, Dosage, and Warning. (n.d.). Retrieved from https://www.webmd.com/vitamins/ai/ingredientmono-842/artichoke
- [Background] 3. Chamomile Plant, Tea, and Oils: Health Benefits and Uses. (n.d.). Retrieved from https://www.webmd.com/diet/supplement-guide-chamomile#1
- [Background] 5. Dyspepsia (Indigestion). (2011, March 01). Retrieved from https://www.aafp.org/afp/2011/0301/p554.html
- [Background] 6. Friedman, L. M., Furberg, C., DeMets, D. L., Reboussin, D., & Granger, C. B. (2015). Fundamentals of clinical trials. Cham: Springer.
- [Background] Giacosa A, Guido D, Grassi M, Riva A, Morazzoni P, Bombardelli E, Perna S, Faliva MA, Rondanelli M. The Effect of Ginger (Zingiber officinalis) and Artichoke (Cynara cardunculus) Extract Supplementation on Functional Dyspepsia: A Randomised, Double-Blind, and Placebo-Controlled Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:915087. doi: 10.1155/2015/915087. Epub 2015 Apr 14. PMID 25954317
- [Background] 8. Ginger Uses, Benefits & Dosage (n.d.). Retrieved from https://www.drugs.com/npp/ginger.html
- [Background] Holtmann G, Adam B, Haag S, Collet W, Grunewald E, Windeck T. Efficacy of artichoke leaf extract in the treatment of patients with functional dyspepsia: a six-week placebo-controlled, double-blind, multicentre trial. Aliment Pharmacol Ther. 2003 Dec;18(11-12):1099-105. doi: 10.1046/j.1365-2036.2003.01767.x. PMID 14653829
- [Background] 10. Licorice: Uses, Side Effects, Interactions, Dosage, and Warning. (n.d.). Retrieved from https://www.webmd.com/vitamins/ai/ingredientmono-881/licorice
- [Background] 11. Marshmallow: Uses, Side Effects, Interactions, Dosage, and Warning. (n.d.). Retrieved from https://www.webmd.com/vitamins/ai/ingredientmono-774/marshmallow
- [Background] 12. McMahon, G. (2019). Comparison of a Numeric and a Descriptive Pain Scale in the Occupational Medicine Setting. Retrieved from https://scholarworks.sjsu.edu/etd_doctoral/98/
- [Background] 13. The R Project for Statistical Computing. (n.d.). Retrieved from https://www.R-project.org/.
- [Background] 14. Vitamin C. (2017, October 18). Retrieved from https://www.mayoclinic.org/drugs-supplements-vitamin-c/art-20363932
- [Background] Leidy NK, Farup C, Rentz AM, Ganoczy D, Koch KL. Patient-based assessment in dyspepsia: development and validation of Dyspepsia Symptom Severity Index (DSSI). Dig Dis Sci. 2000 Jun;45(6):1172-9. doi: 10.1023/a:1005558204440. PMID 10877234
- [Background] Chandrasekaran CV, Sundarajan K, Gupta A, Srikanth HS, Edwin J, Agarwal A. Evaluation of the genotoxic potential of standardized extract of Glycyrrhiza glabra (GutGard). Regul Toxicol Pharmacol. 2011 Dec;61(3):373-80. doi: 10.1016/j.yrtph.2011.10.002. Epub 2011 Oct 13. PMID 22019788
- [Background] Larkworthy W, Holgate PF. Deglycyrrhizinized liquorice in the treatment of chronic duodenal ulcer. A retrospective endoscopic survey of 32 patients. Practitioner. 1975 Dec;215(1290):787-92. PMID 772652
- [Background] Raveendra KR, Jayachandra, Srinivasa V, Sushma KR, Allan JJ, Goudar KS, Shivaprasad HN, Venkateshwarlu K, Geetharani P, Sushma G, Agarwal A. An Extract of Glycyrrhiza glabra (GutGard) Alleviates Symptoms of Functional Dyspepsia: A Randomized, Double-Blind, Placebo-Controlled Study. Evid Based Complement Alternat Med. 2012;2012:216970. doi: 10.1155/2012/216970. Epub 2011 Jun 16. PMID 21747893
- [Background] 19. Rational Phytotherapy: A Physician's Guide to Herbal Medicine. Schulz V, Hansel R, Tyler VE. Terry C. Telger, transl. 3rd ed. Berlin, GER: Springer, 1998.
- [Background] 20. Marshmallow soothes cough. Bone K. Br J Phytother 1993;3(2):93.
- [Background] 21. Antitussive Activity of a Rhamnogalacturonan Isolated from the Roots of Althaea Officinalis L., Var. Robusta. Gabriela Nosáľvá DMartin, Slovakia , Anna Strapková , Alžbeta Kardošová & Peter Capek Journal of Carbohydrate Chemistry Volume 12, 1993 - Issue 4-5
- [Background] Basch E, Ulbricht C, Hammerness P, Vora M. Marshmallow (Althaea officinalis L.) monograph. J Herb Pharmacother. 2003;3(3):71-81. No abstract available. PMID 15277059
- [Background] Haniadka R, Saldanha E, Sunita V, Palatty PL, Fayad R, Baliga MS. A review of the gastroprotective effects of ginger (Zingiber officinale Roscoe). Food Funct. 2013 Jun;4(6):845-55. doi: 10.1039/c3fo30337c. Epub 2013 Apr 24. PMID 23612703
- [Background] Hu ML, Rayner CK, Wu KL, Chuah SK, Tai WC, Chou YP, Chiu YC, Chiu KW, Hu TH. Effect of ginger on gastric motility and symptoms of functional dyspepsia. World J Gastroenterol. 2011 Jan 7;17(1):105-10. doi: 10.3748/wjg.v17.i1.105. PMID 21218090
- [Background] Saller R, Iten F, Reichling J. [Dyspeptic pain and phytotherapy--a review of traditional and modern herbal drugs]. Forsch Komplementarmed Klass Naturheilkd. 2001 Oct;8(5):263-73. doi: 10.1159/000057236. German. PMID 11694755
- [Background] Villa-Rodriguez JA, Kerimi A, Abranko L, Tumova S, Ford L, Blackburn RS, Rayner C, Williamson G. Acute metabolic actions of the major polyphenols in chamomile: an in vitro mechanistic study on their potential to attenuate postprandial hyperglycaemia. Sci Rep. 2018 Apr 3;8(1):5471. doi: 10.1038/s41598-018-23736-1. PMID 29615674
- [Background] Amsterdam JD, Li Y, Soeller I, Rockwell K, Mao JJ, Shults J. A randomized, double-blind, placebo-controlled trial of oral Matricaria recutita (chamomile) extract therapy for generalized anxiety disorder. J Clin Psychopharmacol. 2009 Aug;29(4):378-82. doi: 10.1097/JCP.0b013e3181ac935c. PMID 19593179
- [Background] 28. Functional dyspepsia in adults retrieved from https://www.uptodate.com/contents/functional-dyspepsia-in-adults#H4244969612

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT04153552/Prot_SAP_ICF_000.pdf